CLINICAL TRIAL: NCT01897610
Title: Randomized, Open-label and Multi-center Clinical Trial to Evaluate the Efficacy and Safety of 'Immuncell-LC Group' and 'Non-treatment Group' in Nexavar Treated Patients for Advanced Hepatocellular Carcinoma
Brief Title: Efficacy and Safety of 'Immuncell-LC Group' and 'Non-treatment Group' in Nexavar Treated Patients for Advanced HCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GC Cell Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILC-IIT-04
Record Dates: First submitted 2013-06-25; First posted 2013-07-12 (Estimated); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: Immuncell-LC, advanced hepatocellular carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (No Intervention): The study subjects randomly assigned to the control group is given Nexavar chemotherapy according to the clinical test plans.
- Immuncell-LC group (Experimental): The study subjects assigned to the test group blood is drawn before minimum 2 weeks in order to manufacture the test drug. Test group is compared its progression free survival rate after baseline by administering Nexavar chemotherapy same as control group with Immuncell-LC (10 times).
  Interventions: Drug: Immuncell-LC

INTERVENTIONS:
Drug: Immuncell-LC — intravenous dripping of 200ml(10^9~2x10^10 lymphocytes/60kg adult) for 1 hour
  Other Names: Activated T lymphocyte
  Arms: Immuncell-LC group

SUMMARY:
"Immuncell-LC" in aspects of therapeutic efficacy and safety when administered with Nexavar to advanced Hepatocellular carcinoma patients when compared with the control group who did not receive administration of the drug.

DETAILED DESCRIPTION:
* primary outcome Compare clinical efficacy of group treated with cell therapeutic Immuncell-LC evaluated by progression free survival with that of untreated group
* secondary outcome compare clinical efficacy of group treated with Immuncell-LC, a drug for treating advanced hepatocellular carcinoma evaluated by overall survival, disease control rate, changes of Alpha Feto Protein(AFP) figures from baseline to the last observation date and that of untreated group and evaluate adverse reactions, clinical pathological tests and its safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have consented to the study by providing signature of self, guardian or legal representative
* The patient is more than 20 and less than 80 years old
* The patient is diagnosed as hepatocellular carcinoma by pathological/radiological test and in the stage of III or IV
* Child-Pugh Score should be A
* ECOG Performance Status (ECOG-PS) is less than 2 or equal to
* Patients who receiving or ready for Nexavar treatment
* Patients who satisfy the following conditions of the blood test and kidney function test

  * Absolute granulocyte count is bigger than 1,000/µL
  * Hemoglobin is bigger than 8.5 g/dL
  * Platelet count is bigger than 5x10^10/L
  * Blood Urea Nitrogen(BUN) or Creatinine 1.5xupper normal limit

Exclusion Criteria:

* Patients who are immune deficient or have a history of auto-immune diseases (Ex. Rheumatoid Arthritism, Systemic Lupus Erythematosus, Vasculitis, Multiple sclerosis, Adolescent Insulin-Dependent Diabetes Mellitus, etc.)
* Patients who have a history of malignant tumors in the recent 5 years prior to the study with the exception of basal cell carcinoma, local prostate cancer, and cervical cancer, liver cancer.
* Patients who had anti-cancer medication before the study with the exception of Nexavar
* Patients who has serious dysfunction in other organs by sub-investigator's opinion
* Patients has serious allergic-history by sub-investigator's opinion
* Patients has serious mental disease sub-investigator's opinion
* Pregnant women, nursing mother of having intention of being pregnant during the study
* Patients who participated in other clinical trial within 4 weeks before this study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-12; Primary Completion 2017-07 (Actual); Study Completion 2017-07-04 (Actual)

PRIMARY OUTCOMES:
To assess progression-free survival (PFS) | up to 2 years
  CT, PET-CT, MRI

SECONDARY OUTCOMES:
To assess the overall survival (OS) | up to 2 years
To evaluate the Disease control rate | up to 2 years
  to determine response rate (CR, PR, SD rate) from the baseline to the late observation date using mRECIST
To assess the changes of Alpha Feto Protein(AFP)figures from baseline to the last observation date | up to 2 years
  analysing the changes of AFP before and after combination Nexavar plus Immuncell-LC
Number of participants with adverse events | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Soon Ho Um, MD, PhD, Principal Investigator — Korea University Anam Hospital
Locations (4):
- South Korea (4):
  - Inha University Hospital, Incheon
  - Yonsei University Health System, Seoul
  - Korea University Anam Hospital, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul

REFERENCES:
- [Background] Di Maio M, De Maio E, Perrone F, Pignata S, Daniele B. Hepatocellular carcinoma: systemic treatments. J Clin Gastroenterol. 2002 Nov-Dec;35(5 Suppl 2):S109-14. doi: 10.1097/00004836-200211002-00007. PMID 12394214
- [Background] Ganne-Carrie N, Trinchet JC. Systemic treatment of hepatocellular carcinoma. Eur J Gastroenterol Hepatol. 2004 Mar;16(3):275-81. doi: 10.1097/00042737-200403000-00005. PMID 15195890
- [Background] Cheng AL, Kang YK, Chen Z, Tsao CJ, Qin S, Kim JS, Luo R, Feng J, Ye S, Yang TS, Xu J, Sun Y, Liang H, Liu J, Wang J, Tak WY, Pan H, Burock K, Zou J, Voliotis D, Guan Z. Efficacy and safety of sorafenib in patients in the Asia-Pacific region with advanced hepatocellular carcinoma: a phase III randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2009 Jan;10(1):25-34. doi: 10.1016/S1470-2045(08)70285-7. Epub 2008 Dec 16. PMID 19095497
- [Background] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Background] Furuse J, Ishii H, Nakachi K, Suzuki E, Shimizu S, Nakajima K. Phase I study of sorafenib in Japanese patients with hepatocellular carcinoma. Cancer Sci. 2008 Jan;99(1):159-65. doi: 10.1111/j.1349-7006.2007.00648.x. Epub 2007 Oct 22. PMID 17953709
- [Background] Shim JH, Park JW, Choi JI, Park BJ, Kim CM. Practical efficacy of sorafenib monotherapy for advanced hepatocellular carcinoma patients in a Hepatitis B virus-endemic area. J Cancer Res Clin Oncol. 2009 Apr;135(4):617-25. doi: 10.1007/s00432-008-0496-x. Epub 2008 Oct 10. PMID 18846384
- [Background] Takayama T, Sekine T, Makuuchi M, Yamasaki S, Kosuge T, Yamamoto J, Shimada K, Sakamoto M, Hirohashi S, Ohashi Y, Kakizoe T. Adoptive immunotherapy to lower postsurgical recurrence rates of hepatocellular carcinoma: a randomised trial. Lancet. 2000 Sep 2;356(9232):802-7. doi: 10.1016/S0140-6736(00)02654-4. PMID 11022927
- [Background] Kim HM, Lim J, Yoon YD, Ahn JM, Kang JS, Lee K, Park SK, Jeong YJ, Kim JM, Han G, Yang KH, Kim YJ, Kim Y, Han SB. Anti-tumor activity of ex vivo expanded cytokine-induced killer cells against human hepatocellular carcinoma. Int Immunopharmacol. 2007 Dec 15;7(13):1793-801. doi: 10.1016/j.intimp.2007.08.007. Epub 2007 Aug 31. PMID 17996690